CLINICAL TRIAL: NCT00373204
Title: Phase II Trial of Motexafin Gadolinium and Docetaxel for Second Line Treatment of Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Study of the Effect on Non-small Cell Lung Cancer of the Investigational Drug Motexafin Gadolinium When Used in Combination With Docetaxel (Taxotere)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0229
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Lung Cancer
Keywords: Advanced non-small cell lung cancer; Non-small cell lung cancer; Lung cancer; Metastatic lung cancer; Second line treatment for advanced lung cancer; Cancer; Advanced lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — motexafin gadolinium

ARMS (1):
- Xcytrin® (motexafin gadolinium) (Experimental)
  Interventions: Drug: Motexafin Gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium — On Day 1 of each 3 week cycle for up to 12 cycles:
  MGd 10 mg/kg infused over approximately 30 to 60 minutes, followed ≥ 30 minutes later by Docetaxel 75 mg/m2 administered IV over approximately 1 hour.
  Other Names: MGd and Docetaxtel

SUMMARY:
The purpose of this study is to determine if the addition of motexafin gadolinium (study drug) to standard treatment with docetaxel will improve the response rate in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
Preclinical and clinical data suggest that MGd has activity in NSCLC and that the combination of MGd and docetaxel may be more effective that docetaxel alone. In this trial, patients will receive 10 mg/kg MGd followed by 75 mg/m2 once every 3 weeks. This dosing regimen was well tolerated in the Phase I dose escalation trial. A Simon 2-stage trial design will be used; if at least 4 out of 39 evaluable patients in the first stage of the trial demonstrate objective clinical response, the study will proceed to Stage 2, where an additional 22 evaluable patients will be enrolled following the same treatment regimen and assessment schedule as in Stage 1. Patients with stable disease, CR, or PR will continue dosing up to 12 cycles and will be followed for response every 6 weeks until PD, death, or end of study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Histologically or cytologically confirmed diagnosis of NSCLC
* Inoperable Stage IIIA, unresectable Stage IIIB or metastatic NSCLC patients who have received 1 prior platinum-based chemotherapy regimen
* Measurable disease per RECIST
* ECOG performance status score of 0 or 1
* Willing and able to provide written informed consent

Exclusion Criteria:

* Laboratory values of: ANC < 1500/mm³, Platelet count < 100,000/mm³, hemoglobin < 10 g/dL, AST or ALT > 2.5 x upper limit of normal (ULN), Alkaline phosphatase > 5 x ULN, bilirubin > 1.5 x ULN, serum creatinine > 2.0 mg/dL (176 umol/dL), albumin < 3.0 g/dL (30 g/L)
* Symptomatic or uncontrolled (untreated or treated and progressing) brain metastases
* Evidence of meningeal metastasis
* > 1 prior cytotoxic regimen (not counting adjuvant or neo-adjuvant cytotoxic chemotherapy if completed > 12 months prior to cytotoxic regimen, or prior MGd)
* Chemotherapy, radiation therapy, experimental therapy, immunotherapy, or systemic biologic anticancer therapy within 21 days before beginning study treatment
* Significant weight loss ≥ 10% of body weight within preceding 6 weeks
* Treatment for another cancer within 3 years before enrollment, except basal cell carcinoma of the skin or cervical cancer in situ
* Myocardial infarction within 6 months of enrollment or congestive heart failure rated New York Heart Association Class III or IV
* Uncontrolled hypertension (systolic blood pressure > 160 mm Hg and diastolic blood pressure > 110 mm Hg on maximal medical therapy)
* Known history of porphyria (testing not required at screening visit)
* Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency (testing not required at screening visit)
* History of hypersensitivity to taxanes or polysorbate 80
* Known history of HIV infection (testing not required at screening visit)
* Female who is pregnant or lactating (serum pregnancy test is required for all female patients of childbearing potential)
* Sexually active male or female of childbearing potential unwilling to use adequate contraceptive protection
* Physical or mental condition that makes patient unable to complete specified follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To assess the complete and partial response rate (CR and PR) in patients with advanced NSCLC when administered motexafin gadolinium (MGd) and docetaxel | up to 12 cycles
  The patient population for the primary endpoint is all patients who underwent at least 1 cycle of treatment and at 1 response evaluation.

SECONDARY OUTCOMES:
To estimate the time of progression | up to 12 cycles
  The progression is defined as the time fromfirst does of MGd to first eviedence of progression
To estimate overall survival | up to 12 cycles
  The patient population for this endpoint is all patients who received at least 1 dose of MGd and docetaxel
To estimate progression-free survival | up to 12 cycles
  Progression-free survival is defined as the time from first does of MGd to the earlier of progression
To estimate duration of response (CR + PR) | Up to 12 cycles
  Duration of response (CR +PR) is defined as the time from the fisrt response to the time of disease progression.
To estimate clinical benefit rate (CR + PR + stable disease [SD]) | up to 12 cycles
  The patient population for this endpoint is all patients who underwent at least 2 cycles of treatment and at least 1 response evaluation
To evaluate the safety and tolerability of the combination of MGd and docetaxel in advanced NSCLC | Up to 12 cycles
  All patients who receive at one dose of MGd will be included in the safety summaries and analyses

CONTACTS AND LOCATIONS:
Overall Officials: Kishan Pandya, MD, Study Chair — University of Rochester, Rochester, NY, USA
Locations (22):
- United States (7):
  - Wilshire Oncology Medical Group, La Verne, California
  - University of Rochester, Rochester, New York
  - Tri-County Hematology & Oncology Associates, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Cancer Specialists of Tidewater, Chesapeake, Virginia
- Canada (3):
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - Hospital Charles Lemoyne, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Russia (8):
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk
  - Blokhin Cancer Research Center (Dept. of Chemotherapy), Moscow
  - Blokhin Cancer Research Center (Dept. of Clinical Pharmacology and Chemotherapy), Moscow
  - Central Clinical Hospital, Moscow
  - Moscow Oncology Hospital #62, Moscow
  - St. Petersburg City Oncology Center, Saint Petersburg
  - Samara Regional Oncology Center, Samara
  - Regional Oncology Dispensary, Yaroslavl
- Serbia (4):
  - Clinic for Pulmonary Diseases, Military Medical Academy, Belgrade
  - Clinic for Pulmonary Diseases, Belgrade
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz